CLINICAL TRIAL: NCT01227447
Title: Investigation of the Suburothelial Myofibroblast Network and of Smooth Muscle Function and Control in the Continent and Incontinent Human Urinary Outflow Tract
Brief Title: Investigation of the Suburothelial Myofibroblast Network and of Smooth Muscle Function and Control in the Human Urinary Outflow Tract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Alexander Roosen, PD Dr A Roosen, Ludwig-Maximilians - University of Munich
Other Study IDs: RO 3589/2-1
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Incontinence, Overactive Bladder, Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Stress

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Human tissue from the urinary outflow tract (bladder base and urethra) of patients undergoing cystectomy or radical prostatectomy (for cancer treatment) with pre-operatively documented voiding disorders/incontinence - in particular SUI
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim is to find out if adreno-muscarinic synergy is present also in human tissues of the urinary outflow tract that have a dual adrenergic-muscarinic receptor fitting. To further characterise morphology and function of the suburothelial myofibroblast network in the human bladder outlet.

ELIGIBILITY:
Inclusion Criteria:

Tissue will be collected from the operation theatre only after having obtained the patient´s consent and in strictest accordance with histopathological requirements, i.e. after assessment of resection margins. It might be necessary to retrieve the tissue from the pathologist after first pathological assessment is completed. Tissue will be placed in Tyrode´s solution, gassed with 95 % O2 and 5 % CO2, for functional and RT-PCR or Western blot experiments, or in OCT (optimal cutting temperature) compound, snap-frozen in liquid nitrogen, and stored in a -80°C freezer until cutting for immunohistochemical experiments.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Human tissue from the urinary outflow tract (bladder base and urethra) of patients undergoing cystectomy or radical prostatectomy (for cancer treatment) with pre-operatively documented voiding disorders/incontinence - in particular SUI
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Roosen, PD Dr, Principal Investigator — LMU Munich
Locations (1):
- Ludwig Maximilians University Munich, Dep Urology, Munich, Germany

REFERENCES:
- [Derived] Walther S, Strittmatter F, Hennenberg M, Gratzke C, Stief CG, Roosen A. Adreno-muscarinic synergy in the male human urinary outflow tract. Neurourol Urodyn. 2018 Sep;37(7):2128-2134. doi: 10.1002/nau.23578. Epub 2018 Apr 20. PMID 29675856